CLINICAL TRIAL: NCT01066143
Title: Pharmacotherapy of Generalized Anxiety Disorder With Seroquel: Normalization of Brain Stress and Reward Function
Brief Title: Generalized Anxiety and Seroquel
Acronym: GAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The underwriter stopped the funding
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Igor Elman, MD, MD, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-001662
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Generalized Anxiety Disorder; Seroquel XR
Keywords: Seroquel; Generalized Anxiety Disorder; fMRI
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Seroquel XR (Experimental)
  Interventions: Drug: Seroquel XR

INTERVENTIONS:
Drug: Seroquel XR — Seroquel XR tablets will be flexibly dosed and begun at a target dose of 50 mg on day 1, 100 mg on day 2, 150 mg on day 3 and 200 mg on day 4 with a maximal daily dose of 400 mg on subsequent days.

SUMMARY:
The 12 week clinical trial of Seroquel in Generalized Anxiety Disorder (GAD) patients will be combined with fMRI experiments.

DETAILED DESCRIPTION:
Subjects will be recruited from clinic patients and known research subjects at McLean Hospital, as well as by advertisements in the media, flyers, and word of mouth. An initial telephone interview will be conducted to determine if potential subjects meet the basic study requirements. Subjects will be also screened for drug use. If no obvious health problems are present, subjects will be scheduled for an evaluation. Upon arrival at the research unit, each subject will first complete a standardized interview schedule designed to obtain personal and background data such as age, marital status, socio-economic status, education, employment, etc. The Research Assistant will give subjects both verbal and written descriptions of the study procedures. After briefing subjects on the reasons for the research, subjects will be given the opportunity to ask questions. When they are ready, subjects will be asked to sign the written informed consent form approved by the Mclean Institutional Review Board (IRB). Functional magnetic resonance imaging scans to examine brain functioning will be obtained from GAD patients (N=30) at baseline and after 12 weeks. Seroquel XR tablets will be flexibly dosed and begun at a target dose of 50 mg on day 1, 100 mg on day 2, 150 mg on day 3 and 200 mg on day 4 with a maximal daily dose of 400 mg on subsequent days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Fluency in English
* A diagnosis of GAD
* No pregnancy
* Right-handedness
* Psychotropic medication-free at the start of the study

Exclusion Criteria:

* Pregnancy or lactation
* Any current DSM-IV-TR Axis I disorder
* Any mental retardation or cognitive impairment that precludes informed consent
* Known intolerance or lack of response to quetiapine fumarate
* Substance or alcohol dependence at enrollment
* Participation in another drug trial within 4 weeks prior enrollment
* History of allergic reaction or hypersensitivity to Seroquel or Seroquel XR
* History of prior Seroquel or other antipsychotic agents use
* Contraindications to magnetic resonance imaging
* Treatment with an effective medication for GAD

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 subjects participated in screening but later were found to be ineligible for study participation
Period: Overall Study
Arm/Group | Seroquel XR
Started | 8
Completed | 0
Not Completed | 8
Not completed — ineligible for the study | 8

BASELINE CHARACTERISTICS:
Population: 8 subjects signed the consent but were later found to be ineligible; therefore the study didn't start
Arm/Group | Seroquel XR
Number analyzed (Participants) | 0
Age, Categorical — 8 subjects signed the consent but were later found to be ineligible
  value
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male — 8 subjects signed the consent but were later found to be ineligible
  value
    Female | 0
    Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in GAD Symptomatology at the Week 12 Timepoint.
Description: Changes in anxiety symptomatolgy
Time Frame: 12 week
Population: 8 subjects signed the consent but were later found to be ineligible; the study didn't start
Arm/Group | Seroquel XR
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Time Frame: No adverse events collected. 8 subjects signed the consent but were later found to be ineligible; the study didn't start
Description: 8 subjects signed the consent but were later found to be ineligible; the study didn't start
Arm/Group | Seroquel XR
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
8 subjects signed the consent but were later found to be ineligible; the study didn't start

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes